CLINICAL TRIAL: NCT06963333
Title: Clinical Study on Improving Exercise Capacity in Chronic Obstructive Pulmonary Disease Through Smart IoT-Remote Home Breathing Guidance: A Multicenter, Randomized, Controlled Clinical Trial
Brief Title: Clinical Study on Improving Exercise Capacity in Chronic Obstructive Pulmonary Disease Through Smart IoT-Remote Home Breathing Guidance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Collaborators: Shanxi Bethune Hospital (Other); Henan Fantasy Intelligent Technology Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Daoyin for COPD
Record Dates: First submitted 2025-04-17; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Stable stage of chronic obstructive pulmonary disease; Tele-home rehabilitation; randomized controlled trial
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Breathing guided rehabilitation group (Experimental): The breathing guided rehabilitation group will receive conventional western medicine treatment and breathing guided exercise which consists of training and patient education. They will be evaluated with some tests for the study.
  Interventions: Behavioral: Breathing guided exercise
- Flat ground walking training (Active Comparator): The flat ground walking training group will receive conventional western medicine treatment and flat walking training which consists of training and patient education. They will be evaluated with some tests for the study.
  Interventions: Behavioral: Flat walking training

INTERVENTIONS:
Behavioral: Breathing guided exercise — Breathing guided exercise are divided into six sections: relaxing standing, two fields breathing, regulating lung and kidney, turning side finger, running kidney hall and nourishing qi and collecting gong. Exercise time: 5 days a week, 1 to 2 times a day, a total of 24 weeks.
  Arms: Breathing guided rehabilitation group
Behavioral: Flat walking training — Flat walking training can be performed either outdoors or on flat indoor surfaces at a steady pace of 80 to 120 steps per minute for at least 30 minutes each session, raising the heart rate to the target range and maintaining it for over 10 minutes. This should be done 3 to 5 times a week, with 1 to 2 sessions each day, for a total of 24 weeks. The intensity of the exercise is moderate. The target heart rate based on heart rate reserve is calculated as (maximum heart rate during exercise - resting heart rate) × (40-60)% + resting heart rate.
  Arms: Flat ground walking training

SUMMARY:
This study aims to evaluate the clinical efficacy of breath-guided improvement of COPD exercise ability, establish a breath-guided rehabilitation program of intelligent iot and remote home, improve COPD exercise ability, reduce acute exacerbation, and form high-quality clinical evidence.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is the most common chronic airway disease in China. Based on the digital management platform, 548 patients with COPD in stable stage were selected as the research objects. A multi-center, randomized, controlled clinical trial design was adopted to scientifically evaluate the clinical efficacy of breath-guided improvement of COPD exercise ability and reveal its mechanism of action. A breath-guided rehabilitation program based on intelligent iot and remote home was established and promoted to improve exercise ability and reduce acute exacerbation. To form high-quality clinical evidence, and realize tracking management, real-time evaluation and effect evaluation throughout rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD in stable stage
* Patients with grade 2 to 4 lung function
* Age 40~80 years old
* Be able to use smart phones, computers and other devices independently or with the help of family members during home training
* Volunteer for treatment and sign an informed consent form

Exclusion Criteria:

* Pregnant or lactating women and patients with recent pregnancy plans
* Delirious, dementia, all kinds of mental illness
* Tumor patients who have undergone resection, radiation, and chemotherapy within 5 years
* Patients with severe osteoarthropathy or osteoporosis, unstable fractures
* Patients with severe visual impairment that cannot be improved or who have epilepsy or vertigo and cannot use VR devices
* Patients with progressive neuromuscular disease
* Patients with pulmonary abscess, pulmonary interstitial fibrosis, active pulmonary tuberculosis, bronchiectasis, pulmonary embolism and other pulmonary diseases
* Patients with severe cardiovascular and cerebrovascular diseases (malignant arrhythmia, unstable angina pectoris, acute myocardial infarction, grade 3 or above cardiac function, stroke, cerebral hemorrhage, etc.)
* Patients with severe liver disease (cirrhosis, portal hypertension and bleeding caused by esophageal and gastric varices, etc.) and severe kidney disease (dialysis, kidney transplantation, etc.)
* Participants who were participating in other clinical trials within 1 month prior to enrollment
* People who stay in bed for a long time for various reasons

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 548 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
6 Minutes Walking Distance Test (6MWD) | Changes in baseline 6MWD test at weeks 12 and 24 of the treatment period and at 28 weeks of follow-up.
  The 6-minute walking distance of the two groups was calculated

SECONDARY OUTCOMES:
Incidence of acute exacerbation | Changes in baseline Incidence of acute exacerbation at weeks 12 and 24 of the treatment period and at 28 weeks of follow-up.
  The proportion of patients with ≥1 acute exacerbation in each group during the study period was recorded. If the interval between two acute exacerbations was within 5 days, it was considered as 1 acute exacerbation.
Degree of breathing difficulty | Changes in baseline mMRC scores at weeks 12 and 24 of the treatment period and at 28 weeks of follow-up.
  The modified Medical Research Council dyspnoea scale (mMRC) will be used to assess severity of dyspnea. The mMRC scale is a 4-point (0-4) scale. "0" means no dyspnea perception, "4" means severe dyspnea perception.
Borg dyspnea score | Changes in baseline Borg dyspnea score at weeks 12 and 24 of the treatment period and at 28 weeks of follow-up.
  Borg dyspnea score is a 10-point (0-10) scale based on the severity of dyspnoea. "0" means no dyspnea perception, "10" means most severe dyspnea perception.
The COPD Assessment Test(CAT) | Changes in baseline CAT scores at weeks 12 and 24 of the treatment period and at 28 weeks of follow-up.
  The COPD Assessment Test (CAT) is an 8-item questionnaire that assesses health status in patients with COPD. The questionnaire uses a 0-5 point scale, with higher values indicating a greater impact of COPD on the patient.
Lung function | Changes in baseline Lung function test at weeks 0 and 24 of the treatment.
  Forced Vital Capacity (FVC)、Forced Expiratory Volume in One Second (FEV1) and Percentage of Forced Expiratory Volume in One Second to Predicted Value (FEV1% pred) were mainly used for lung function evaluation.
Anxiety Scale | Changes in baseline SAS scores at weeks 12 and 24 of the treatment period and at 28 weeks of follow-up.
  The Self-Rating Anxiety Scale (SAS) was used to assess the anxiety state of patients. It is a questionnaire consisting of 20 items, with a score range of 1 to 4. The higher the value, the more severe the anxiety state of the patients.
Depression Scale | Changes in baseline SDS scores at weeks 12 and 24 of the treatment period and at 28 weeks of follow-up.
  The Self-Rating Depression Scale (SDS) was used to assess the depressive state of patients. It is a questionnaire consisting of 20 items, with a score range of 1 to 4. The higher the value, the more severe the depressive state of the patients.
Clinical symptom assessment questionnaire (CCQ) | Changes in baseline CCQ scores at weeks 12 and 24 of the treatment period and at 28 weeks of follow-up.
  The Clinical symptom assessment questionnaire (CCQ) is a self-administered questionnaire that measures healthrelated quality of life. It is an 10-item questionnaire on a 0-6 point scale with higher values indicating greater impact of COPD.
St. George's Respiratory Questionnaire (SGRQ) | Changes in baseline SGRQ scores at weeks 12 and 24 of the treatment period and at 28 weeks of follow-up.
  The St. George's Respiratory Questionnaire (SGRQ) scores will be used to evaluate quality of life with a total score of 0-100. The higher scores will indicate the worse outcomes.
The modified Effectiveness Satisfaction Questionnaire for COPD (mESQ-COPD) | Changes in baseline mESQ-COPD scores at weeks 12 and 24 of the treatment period and at 28 weeks of follow-up.
  The modified Effectiveness Satisfaction Questionnaire for COPD (mESQ-COPD) will be used to assess treatment satisfaction. The mESQ-COPD contains 19 items in four domains. mESQ-COPD scores range from 0 to 4 with a decrease in score showing higher treatment satisfaction.
The modified COPD Patient-Reported Outcome scale (mCOPD-PRO) | Changes in baseline mCOPD-PRO scores at weeks 12 and 24 of the treatment period and at 28 weeks of follow-up.
  The modified COPD Patient-Reported Outcome scale (mCOPD-PRO) will be used to assess quality of life. The mCOPD-PRO contains 27 items in three domains. mCOPD-PRO scores range from 0 to 4 with a decrease in score showing higher health status.

CONTACTS AND LOCATIONS:
Overall Officials: Jiansheng Li, doctor, Study Chair — The First Affiliated Hospital of Henan University of Traditional Chinese Medicine
Locations (1):
- The First Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan, China